CLINICAL TRIAL: NCT05414838
Title: Pilot Assessment of the Safety of a Combination of Curcumin, Omega-3, and Vitamin D Supplements (PASCOD) in Healthy Human Volunteers
Brief Title: Pilot Assessment of the Safety of a Combination of Curcumin, Omega-3, and Vitamin D Supplements
Acronym: PASCOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH1-168004
Record Dates: First submitted 2022-05-09; First posted 2022-06-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-05

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Curcumin; Docosahexaenoic Acids; Cholecalciferol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Curcumin, Omega-3 and Vitamin-D (COD) (Experimental)
  Interventions: Dietary Supplement: Curcumin, Omega-3 and Vitamin-D (COD)

INTERVENTIONS:
Dietary Supplement: Curcumin, Omega-3 and Vitamin-D (COD) — Acumin™ Turmeric Complex (Dr. D's Ultra BioTurmeric) 500 mg daily (NPN 80087842)
  Omega-3 supplements (combination of DHA and EPA) 900 mg daily (NPN 80019234)
  Vitamin D3 supplements 2500 IU daily (NPN 80108995)

SUMMARY:
Curcumin, Omega-3 and Vitamin-D (COD) are commonly used dietary supplements, which are licensed natural health products in Canada. The investigators are interested to see what effects (good or bad) these supplements taken in combination, might have on a person and the potential impact of these supplements, in combination, on inflammation and the immune system, in the body. This is because the investigators study Rheumatoid Arthritis (RA), an autoimmune disease that affects the joints of the body, causing joint pain and swelling.

The investigators want to first evaluate the tolerability and potential negative effects of these three supplements in combination, also known as "side-effects" in healthy persons. This pilot study will also help us determine the length of time research participants need for their research visits for future clinical trials.

The investigators also want to explore the utility and validity of two different 24-hour food recall methods (ASA24-Canada-2018 and Keenoa food diary) and the dietary inflammatory index (DII) using both recall methods. The DII is a score calculated from dietary data, to establish the inflammatory potential of an individual's diet.

This research pilot study aims to enroll 50 persons. The investigators want to identify common side effects of the supplements when all three are taken together, as well as any other potential side-effects that might occur that are not common. Based on the scientific research, persons who have taken these supplements individually (e.g., Vitamin D alone or Omega-3 alone), show that serious side effects are unlikely and if they do occur are mild. Pure curcumin, like that being administered in this study, containing no fillers, has not shown to have adverse effects and is well tolerated. However, no scientific studies have been done using all three of these nutritional supplements together, in humans.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give free informed consent and written consent in English, for participation in the trial
* Participant will provide contact information that includes telephone, email address and mailing address
* Age between 18 and 49 years old
* BMI range between 18.5 - 34.9 (kg/m2)
* Female participants of child-bearing potential must be willing to ensure that they use effective contraception during the trial
* Participant has clinically acceptable laboratory results including routine hematology (CBC) and biochemistry (electrolytes, creatinine, ALT, ALP, GGT, AST, Glucose)
* In the Investigator's opinion, is able and willing to comply with all trial requirements
* Participant is an employee or student at the Health Sciences Centre or Bannatyne Campus, by self-report
* Participants currently taking vitamin D and/or omega-3 supplements are willing to stop taking their own supplements prior to the start of this trial.
* Participant has received two-doses of a COVID-19 vaccine, with the second dose occurring no less than 4 weeks before Visit 1

Exclusion Criteria:

* Any history of clinically important and poorly controlled autoimmune disorders, endocrine disorders, cardiovascular disease, pulmonary, biliary or GI disorders, or any history of cancer requiring chemotherapy or radiation within the last 1 year
* Current use of warfarin or similar anticoagulant medication (at the discretion of the P.I.)
* Stomach ulcers (e.g., active peptic ulcer disease within the last 6 weeks) or poorly controlled gastric esophageal reflux disease (GERD)
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
* Female of childbearing potential who is unwilling to ensure effective contraception during the trial
* Scheduled elective surgery or other procedures requiring general anesthesia during the trial
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Concurrent commitment to enroll in another clinical trial
* Regular daily consumption of a Curcumin containing product within the last three months
* Self-report of allergic reaction to fish
* Self-reported body weight change of greater than 3.5 kg within the past 3 months, unexplained by medical history
* Participants who indicate that they will not consume the treatments on a daily basis
* Recent history (within 12 months of screening) or current consumption of > 14 drinks per week, (1 drink = 12oz of beer, 5oz of wine or 1.5oz distilled spirits)
* Participants who report they have had viral or bacterial infection in the last 4 weeks (e.g.COVID-19, the flu, a cold, stomach flu, bladder infection, strep throat), and are not fully recovered
* Participants who have been vaccinated in the last 4 weeks and in the opinion of the Investigator may influence the result of the trial.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Self-reported Side Effects due to Supplements | 4 weeks
  Participants will fill out a weekly monitoring survey to report side effects and health issues they may have had over the past week while taking the COD supplements. Participants will fill out a short survey weekly using a 0-3 scale of severity for a variety of gastrointestinal and health symptoms to analyze total side effects over the trial.

SECONDARY OUTCOMES:
Supplementation adherence | Day 28
  Medication adherence (>75% pills consumed) Non-adherence (<75% of the capsules consumed)
  Medication packs will be returned on Day 28 (+/- 2 days) of the trial. Remaining capsules will be counted and deemed to have been missed.

OTHER OUTCOMES:
Alanine transaminase (ALT) | Baseline, Day 28
  ALT is measured in U/L
Aspartate Aminotransferase (AST) | Baseline, Day 28
  AST is measured in U/L
Alkaline Phosphatase (ALK) | Baseline, Day 28
  AST is measured in U/L
Total Bilirubin | Baseline, Day 28
  Total blood bilirubin is measured in μmol/L
Direct Bilirubin | Baseline, Day 28
  Direct bilirubin is measured in μmol/L
Urea | Baseline, Day 28
  The total blood urea concentration in mmol/L
Glucose | Baseline, Day 28
  Total fasted blood glucose concentration in mmol/L
Total Cholesterol | Baseline, Day 28
  Total cholesterol measured in mmol/L
Low-density lipoprotein (LDL) | Baseline, Day 28
  LDL measured in mmol/L
High-density lipoprotein (HDL) | Baseline, Day 28
  HDL measured in mmol/L
Triglycerides | Baseline, Day 28
  Non-fasted triglycerides measured in mmol/L
Sodium | Baseline, Day 28
  Total blood sodium concentration in mmol/L
Potassium | Baseline, Day 28
  Total blood potassium concentration in mmol/L
Chloride | Baseline, Day 28
  Total blood chloride concentration in mmol/L
Calcium | Baseline, Day 28
  Total blood calcium concentration in mmol/L
Bicarbonate | Baseline, Day 28
  Bicarbonate measured in mmol/L
Magnesium | Baseline, Day 28
  Magnesium measured in mmol/L
Albumin | Baseline, Day 28
  Total blood albumin concentration in g/L
Phosphate | Baseline, Day 28
  Total blood phosphate concentration in mmol/L
Creatinine | Baseline, Day 28
  Total blood creatinine concentration in μmol/L
C-Reactive Protein (CRP) | Baseline, Day 28
  CRP measured in mg/L
White blood cells (WBC) | Baseline, Day 28
  WBC measured in x10^9/L
Hemoglobin | Baseline, Day 28
  Hemoglobin measured in g/L
Platelets | Baseline, Day 28
  Platelets measured in x10^9/L
Mean platelet volume (MVP) | Baseline, Day 28
  MVP measured in fL
Body weight | Baseline, Day 28
  Body weight will be measured in kg
Waist circumference | Baseline, Day 28
  Waist circumference will be measured in cm
Systolic Blood Pressure | Baseline, Day 28
  Systolic blood pressure in mmHg
Diastolic Blood Pressure | Baseline, Day 28
  Diastolic blood pressure in mmHg
Hand Grip Strength | Baseline, Day 28
  Measured using a dynamometer in kg, taken in triplicate
Tender and Swollen Joint Count (TSJC) | Baseline, Day 28
  44 joints assessed by a rheumatologist
Physician Global Assessment of Disease Activity | Baseline, Day 28
  Severity measured on a scale from 0 to 10
Routine Assessment of Patient Index Data 3 (RAPID 3) | Baseline, Day 28
  Disease activity index calculated from a short and questionnaire
Simple Disease Activity Index (SDAI) | Baseline, Day 28
  A score that determines severity of rheumatoid arthritis using clinical and laboratory data
Clinical Disease Activity Index (CDAI) | Baseline, Day 28
  A score that determines severity of rheumatoid arthritis using only clinical data
Disease Activity Score-28- C-Reactive Protein (DAS28-CRP) | Baseline, Day 28
  A score that describes severity of rheumatoid arthritis using clinical data and CRP
Dietary Inflammatory Index | Baseline, Day 28
  A score calculated from dietary data, to establish the inflammatory potential of an individual's diet.

CONTACTS AND LOCATIONS:
Overall Officials: Liam O'Neil, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada